CLINICAL TRIAL: NCT02261428
Title: Randomized Controlled Study of Nasotracheal Suction With Tiemann Catheter Compared to the Classic Technique With the Standard One.
Brief Title: Nasotracheal Suction With Tiemann Catheter Compared to the Classic Technique With the Suction Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grigoriadis Konstantinos (Other)
Responsible Party: Sponsor-Investigator, Grigoriadis Konstantinos, Physical Therapist, Attikon Hospital
Organization: Attikon Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: AttikonH
Record Dates: First submitted 2014-09-30; First posted 2014-10-10 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Muscle Weakness
Keywords: Nasotracheal suction, tracheal access
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Catheter Tiemann (Experimental): We tested the ability of Tiemman catheter to access trachea and aspirate bronchial secretions, measuring number of attempts and time required for the intervention
  Interventions: Device: Catheter Tiemann
- Suction catheter (Active Comparator): We tested the ability of suction catheter to access trachea and aspirate bronchial secretions, measuring number of attempts and time required for the intervention
  Interventions: Device: Suction catheter

INTERVENTIONS:
Device: Catheter Tiemann — We tested the ability of Tiemann catheter to access trachea in order to aspirate bronchial secretions in ICU patients
  Arms: Catheter Tiemann
Device: Suction catheter — We tested the ability of Suction catheter to access trachea in order to aspirate bronchial secretions in ICU patients
  Arms: Suction catheter

SUMMARY:
The study compares the effectiveness of Tiemann and Suction catheters, with regard to attempts to enter the trachea and the time required for the procedure.

DETAILED DESCRIPTION:
The population of the study was twenty (20) patients, hospitalized in General and Cardiothoracic ICU, mostly with respiratory failure of various etiologies, the majority of which has complicated with Unit Myoneuropathy. This state confirmed by medical research council (MRC) Sum score which gave a result less than 48/6011 which corresponds to thirteen (13) patients in the total population of the study.

The randomization of the study achieved using the sealed envelopes method and associated with the catheter to be first used in the suction9,10 (Tiemann or suction catheter).

Twenty (20) sealed envelopes were prepared from a team not related to the study. The sealed envelopes had an inside paper with the sign "T" for the first ten (10) envelopes and "N" for the rest ten (10) of them.

When a new patient met the criteria for this study, one sealed envelope was randomly selected to determine the technique would come first: "T" for Tiemann technique or "N" for Suction catheter technique.

Furthermore the following parameters tabulated for each patient:

* Sex
* Unit
* Cause input
* First catheter used
* Second catheter used
* Hospitalization day
* Age
* Possible causes weakness
* Percentage oxygen mixture fraction of inspired oxygen (FiO2) and
* Oxygen partial pressure (PaO2) before any action

In addition to the above, all the parameters needed for calculating the Sequential Organ Failure Assessment score (SOFA) were tabulated, such as:

* Bilirubin
* The Glasgow Coma Score
* Platelets
* Mean arterial pressure
* Creatinine and urine 24 hours

Finally, it was recorded for each patient before and after the two catheterizations as indicators of disturbance and physiological burden attached to the intervention:

* The systolic and diastolic blood pressure
* The respiratory rate
* The heart rate
* The saturation of hemoglobin
* The blood gases, which recorded the partial pressure of oxygen (PaO2), carbon dioxide carbon dioxide partial pressure (PaCO2), the Ph and bicarbonates (HCO3).

A first check took place to identify each patient who met the admission criteria for the study.

The procedure required two people skilled in the nasotracheal suction (NTS), the first one to perform the NTS and the other one to record the time and the attempts needed, and it was beginning by correcting the posture of each patient on the bed, when the Great Trochanter was more than 20 centimeters away from the hinge of the bed.

The pillow beneath the patient's head was removed to have an extended position, the first blood gas analysis was done and the parameters mentioned above were recorded in the relevant tables.

To determine the access of the trachea, it was used a stethoscope to hear turbulent flow on the anterior surface of the chest.

The whole procedure comprises two "steps":

a) Achieving of the entrance into the nasopharynx b) Achieving of the entrance into the trachea

1. To achieve the entrance into the nasopharynx:

   * It was selected the opposite nostril that Levine was placed.
   * The insertion of the catheter was always opposite to the medial canthus of the eye.
   * If it was found resistance and the catheter was not inserted to the nasopharynx, it was pulled slightly outwardly and then inwardly.

   Each kind of micromanipulation recorded as attempt. The maximum number of attempts were agreed in Protocol Design (beyond which the attempts would stop) was five (5). In fact, in no cases was exceeded the limit of five attempts.

   The time recorded corresponds to the time needed for the successful advancement of the catheter in the nasopharynx through the nostril (T1).
2. Achieving of the entrance into the trachea:

The successful insertion of the catheter into the trachea was confirmed by another member of the team using stethoscope and was determined by:

i. Hearing of turbulent flow when closing the "fingertip" ii. Insertion without resistance iii. Tickly cough during the insertion.

The insertion to trachea was considered to be unsuccessful as the catheter insert into the esophagus and thus:

i. There was no production of turbulent airflow when the hole of "fingertip"was closed ii. It was found resistance during the insertion of the catheter iii. There was a grimace of disgust on the patient's face. As the insertion was considered to be unsuccessful according to the above conditions, catheter was drawn slightly outward (less than one centimeter) and redirected to the trachea.

Each kind of micromanipulation recorded as attempt. The maximum number of attempts were agreed in Protocol Design was ten (10). Beyond the above limit the insertion was considered to be unsuccessful and repeated after half an hour15 with the other catheter (half an hour is the sufficient time for the patient to return to his initial condition).

The time of the second "step" recorded, corresponds to the time needed for the successful promotion of the catheter from the nasopharynx to the trachea (T2).

Finally it was recorded the time needed for each suction which was tabulated below as (T3).

The summation of (T1), (T2) and (T3) was reflected the total time needed for the whole procedure which was followed by a new blood gas analysis.

All parameters were recorded by the team involved to the study. The catheters used for this study were 14 French dia. of the same industry and from the same material (medical PVC).

As it was mentioned above, the whole idea based on the J-shape of the Tiemann catheter which is useful for the orientation of the catheter during the insertion to the nasopharynx first and then into the trachea and placed always downwards.

The oxygen face mask was maintained during the insertion of the catheter in order to continue the patient's oxygenation and avoid hypoxemia. This was achieved by leaving outside the oxygen face mask only the opposite nostril of the nasogastric tube.

No extra oxygen was given to patients before the procedure as pre-oxygenation.

The size of the sample was calculated based on a pilot study and was determined to twenty (20) patients were not included in the main study. Thus ten (10) patients underwent an equal number of nasotracheal suctioning with Tiemann catheter and ten (10) with Suction catheter.

For standard deviation σ1=3.9, and an error α=0,05 and power 80, the sample size must be bigger than twelve (12).

From all the above the investigators summarize that the sample size of twenty (20) patients was adequate.

For the statistical analysis was used the SPSS 20 Inc., Chicago, IL, and for paired values the Paired T-Test and Wilcoxon Signed Rank Test.

For paired nominal parameters was used the McNemar Χ2 test. To determine normal distributions, was used the Kolmogorov-Smirnov test. In the majority of cases data are presented as Median (Range) in abnormal distributions and Mean (SD) in normal.

Odds ratio was used to quantify how strongly Tiemann associated with Suction catheter in total attempts.

Significance was taken as P < 0.05. To determine the difference in time needed by using the two catheters was used Kaplan-Mayer analysis and long-rank test.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients with nasogastric tube and spontaneous breathing without artificial airway
* Inability to mobilize and handle secretions
* Glasgow Coma Scale (GCS) >12/15
* PaO2/FiO2 ratio >100

Exclusion Criteria:

* Active nasal bleeding
* international normalized ratio (INR)>3
* Glasgow Coma Scale (GCS) <11/15
* Facial or basal cranial fractures
* Tumor in trachea
* Pregnancy
* ICU patients with endotracheal tube or tracheostomy tube

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Angouras, MD, Study Director — Athens University School of Medicine, Department of Cardiothoracic Surgery; Theodoros Xanthos, MD, Study Director — Athens University School of Medicine, Postgraduate program in CPR (moderator); Konstantinos Grigoriadis, PT, Principal Investigator — Attikon Hospital; Katerina Flevari, MD, Study Chair — Attikon Hospital

REFERENCES:
- [Background] Pode D, Manny J. A simplified method for repeated nasotracheal suction. Surg Gynecol Obstet. 1984 Aug;159(2):173-4. PMID 6463830
- [Background] Brucia J, Rudy E. The effect of suction catheter insertion and tracheal stimulation in adults with severe brain injury. Heart Lung. 1996 Jul-Aug;25(4):295-303. doi: 10.1016/s0147-9563(96)80065-3. PMID 8836745
- [Background] Gemma M, Tommasino C, Cerri M, Giannotti A, Piazzi B, Borghi T. Intracranial effects of endotracheal suctioning in the acute phase of head injury. J Neurosurg Anesthesiol. 2002 Jan;14(1):50-4. doi: 10.1097/00008506-200201000-00010. PMID 11773824
- [Background] Marlow TJ, Goltra DD Jr, Schabel SI. Intracranial placement of a nasotracheal tube after facial fracture: a rare complication. J Emerg Med. 1997 Mar-Apr;15(2):187-91. doi: 10.1016/s0736-4679(96)00356-3. PMID 9144060
- [Background] Sloan EP, VanRooyen MJ. Suction catheter-assisted nasotracheal intubation. Acad Emerg Med. 1994 Jul-Aug;1(4):388-90. doi: 10.1111/j.1553-2712.1994.tb02651.x. PMID 7614287
- [Background] Roppolo LP, Vilke GM, Chan TC, Krishel S, Hayden SR, Rosen P, Trione M. Nasotracheal intubation in the emergency department, revisited. J Emerg Med. 1999 Sep-Oct;17(5):791-9. doi: 10.1016/s0736-4679(99)00085-2. PMID 10499691
- [Background] Saissy JM, Boussignac G, Cheptel E, Rouvin B, Fontaine D, Bargues L, Levecque JP, Michel A, Brochard L. Efficacy of continuous insufflation of oxygen combined with active cardiac compression-decompression during out-of-hospital cardiorespiratory arrest. Anesthesiology. 2000 Jun;92(6):1523-30. doi: 10.1097/00000542-200006000-00007. PMID 10839900
- [Derived] Grigoriadis KEpsilon, Angouras DC, Flevari A, Xathos T. Comparison of the Feasibility and Safety of Nasotracheal Suctioning With Curved Edge Catheter Versus Conventional Suction Catheter in Critically Ill Subjects: A Prospective Randomized Crossover Trial. Respir Care. 2015 Dec;60(12):1826-33. doi: 10.4187/respcare.03875. Epub 2015 Oct 20. PMID 26487746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All ICU patients were breathing spontaneously, had respiratory failure of various pathophysiological mechanisms, with impaired cough reflex
Pre-assignment Details: Of the 30 patients screened during the run-in period between May 2014 and September 2014 they received nasotracheal suction all. 10 of them required for pilot study and 20 for the main study. The pilot study was designated as a separate study and the participants was not included in this record.
Groups:
- Catheter Tiemann First, Then Suction Catheter: Participants first received nasotracheal suction with catheter Tiemann. After a washout period minimum of half hour they received a second nasotracheal suction with Suction catheter
- Suction Catheter First, Then Catheter Tiemann: Participants first received nasotracheal suction with suction catheter. After a washout period minimum of half hour they received a second nasotracheal suction with catheter Tiemann.
Period: Overall Study
Arm/Group | Catheter Tiemann First, Then Suction Catheter | Suction Catheter First, Then Catheter Tiemann
Started | 10 (Washout (30 minutes)) | 10 (Washout (30 minutes))
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The participants were non intubated ICU patients who had inadequate cough leading to the inability to mobilize their secretions. The inadequate cough is result of neuromuscular disorders, ICU neuromyopathy, abdominal pain due to surgery and low consiousness due to head injuries.
Groups:
- Suction Catheter First, Then Catheter Tiemann: Participants first received nasotracheal suction with Suction catheter . After a washout period minimum of half hour they received a second nasotracheal suction with catheter Tiemann.
- Total: Total of all reporting groups
Arm/Group | Catheter Tiemann First, Then Suction Catheter | Suction Catheter First, Then Catheter Tiemann | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Number; unit: participants] — Αge categories were defined in order to reflect the age in relation to the sensitivity of the population it invasive interventions
  participants
    <60 years | 1 | 0 | 1
    60-69 years | 2 | 2 | 4
    70-79 years | 3 | 3 | 6
    >80 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants] — Gender determines the behavior of the autonomic nervous system
  Participants
    Female | 5 | 5 | 10
    Male | 5 | 5 | 10
SOFA [Number; unit: participants] — Used to monitor the patient's condition during the stay in the intensive care unit (ICU).
  Both the mean and highest SOFA scores are predictors of outcome. An increase in SOFA score during the first 24 to 48 hours in the ICU provided a mortality rate of at least 50% to 95%. Scores less than 9 give prediction of mortality by 33%, while over 11 may be near or above 95%
  participants
    <4 | 7 | 7 | 14
    6 | 2 | 2 | 4
    9 | 1 | 1 | 2
Hospitalisation day [Number; unit: participants] — Specifies the degree of ICU neuromyopathy associated with weakness cough.
  participants
    < 5 days | 2 | 2 | 4
    ≥ 5 days, < 10 days | 3 | 3 | 6
    ≥ 10 days | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Attempts Before Entering Trachea
Description: We count the required attempts to insert catheter into trachea (number of attempts)
Time Frame: An average of 15 seconds
Measure: Mean (Standard Deviation); unit: Attempts
Groups:
- Catheter Tiemann: The number below represents the mean of attempts made wth catheter Tiemann.
- Suction Catheter: The number below represents the mean of attempts made wth Suction catheter.
Arm/Group | Catheter Tiemann | Suction Catheter
Number analyzed (Participants) | 19 | 19
Attempts | 2.63 (2.24) | 6.79 (3.75)
Statistical Analysis 1: Comparison: Catheter Tiemann vs Suction Catheter; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 3.95, 95% CI 2-sided [1.79 to 8.73]

2. Secondary Outcome: Time to Entering Trachea
Description: We count the required time needed to insert catheter into trachea (seconds).
Time Frame: An average of 15 seconds
Population: The 19 interventions with each catheter was used randomly
Measure: Mean (Standard Deviation); unit: Sec
Groups:
- Catheter Tiemann: The number below represents the mean of time required to insert the trachea wth catheter Tiemann.
- Suction Catheter: The number below represents the mean of time required to insert the trachea wth Suction catheter
Arm/Group | Catheter Tiemann | Suction Catheter
Number analyzed (Participants) | 19 | 19
Sec | 10.05 (10.074) | 20.06 (12.694)

3. Secondary Outcome: Respiratory Rate Immediately After Intervention
Description: Recorded the respiratory rate (breaths per minute), immediately after intervention
Time Frame: Within 2 seconds after catheter withdrawal.
Measure: Mean (Standard Deviation); unit: Βreaths per minute
Groups:
- Catheter Tiemann: The number below represents the mean of respiratory rate recorded immediately after insertion to trachea wth catheter Tiemann.
- Suction Catheter: The number below represents the mean of respiratory rate recorded immediately after insertion to trachea wth Suction catheter
Arm/Group | Catheter Tiemann | Suction Catheter
Number analyzed (Participants) | 19 | 19
Βreaths per minute | 26.37 (7.544) | 25.79 (7.941)

4. Secondary Outcome: Heart Rate Immediately After Intervention
Description: Immediately after each intervention recorded the heart rate (beats per minute).
Time Frame: Within 2 seconds after catheter withdrawal.
Measure: Mean (Standard Deviation); unit: Βeats per minute
Groups:
- Catheter Tiemann: The number below represents the mean of heart rate recorded immediately after insertion to trachea wth catheter Tiemann.
- Suction Catheter: The number below represents the mean of heart rate recorded immediately after insertion to trachea wth Suction catheter
Arm/Group | Catheter Tiemann | Suction Catheter
Number analyzed (Participants) | 19 | 19
Βeats per minute | 87.21 (15.623) | 86.53 (14.013)

5. Secondary Outcome: Systolic Blood Pressure Immediately After Each Intervention
Description: Immediately after each intervention recorded the systolic blood pressure (mmHg).
Time Frame: Within 2 seconds after catheter withdrawal.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Catheter Tiemann: The number below represents the mean of systolic blood pressure recorded immediately after insertion to trachea wth catheter Tiemann.
- Suction Catheter: The number below represents the mean of systolic blood pressure recorded immediately after insertion to trachea wth Suction catheter
Arm/Group | Catheter Tiemann | Suction Catheter
Number analyzed (Participants) | 19 | 19
mmHg | 143.37 (24.703) | 141.32 (19.136)

6. Secondary Outcome: Diastolic Blood Pressure Immediately After Each Intervention
Description: Immediately after each intervention recorded the diastolic blood pressure (mmHg).
Time Frame: Within 2 seconds after catheter withdrawal.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Catheter Tiemann: The number below represents the mean of diastolic blood pressure recorded immediately after insertion to trachea wth catheter Tiemann.
- Suction Catheter: The number below represents the mean of diastolic blood pressure recorded immediately after insertion to trachea wth Suction catheter
Arm/Group | Catheter Tiemann | Suction Catheter
Number analyzed (Participants) | 19 | 19
mmHg | 62.74 (13.482) | 60.32 (11.856)

7. Secondary Outcome: Presence of Blood on Catheter Immediately After Each Intervention
Description: Immediately after each intervention recorded the presence or absence of blood on the catheter (Yes or No).
Time Frame: Within 2 seconds after catheter withdrawal.
Measure: Number; unit: Catheters with presence of blood
Groups:
- Catheter Tiemann: Presence of blood was found on Participants immediately after suctioning with catheter Tiemann
- Suction Catheter: Presence of blood was found on Participants immediately after suctioning with Suction catheter
Arm/Group | Catheter Tiemann | Suction Catheter
Number analyzed (Participants) | 19 | 19
Catheters with presence of blood | 6 | 6

ADVERSE EVENTS:
Time Frame: 5 months
Description: Presence of Blood on Catheter
Groups:
- Catheter Tiemann: Participants received nasotracheal suction with catheter Tiemann.
- Suction Catheter: Participants received nasotracheal suction with Suction catheter
Arm/Group | Catheter Tiemann | Suction Catheter
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter Tiemann (N=20) | Suction Catheter (N=20)
Presence of Blood on Catheter (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes